CLINICAL TRIAL: NCT04662996
Title: Search for Predictive Factors of Resistance to Treatment for Metastatic Castration-resistant Prostate Cancer by Studying the Expression of microRNAs
Acronym: MiR_CPMRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DR200300 _MiR_CPMRC; 2020-A03304-35 (Registry Identifier: ANSM)
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer; Resistance, Disease; MicroRNAs
MeSH Terms: conditions — Prostatic Neoplasms; Disease Resistance | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Intervention: blood sample at inclusion. primary purpose: to better understand resistance mechanisms to prostate cancer treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1- Chemotherapy (Experimental): Intervention : one blood sample is done before beginning chemotherapy as a first treatment line for a metastatic castration resistant prostate cancer
  Interventions: Biological: Blood sample
- 2- Novel Hormonal Agent (Experimental): Intervention : one blood sample is done before beginning a novel hormonal agent (abiraterone, enzalutamide) as a first treatment line for a metastatic castration resistant prostate cancer
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — one blood sample is done before beginning a first treatment line for a metastatic castration resistant prostate cancer

SUMMARY:
Several drugs are available for metastatic castration resistant prostate cancer such as chemotherapy (docetaxel, cabazitaxel) and novel hormonal agents (abiraterone, enzalutamide), in France. The oncologist has to choose between those two type of treatment, without any biological predictor of efficacy for his patient. It is always difficult to choose knowing that 30 to 50% of patients won't benefit from the treatment chosen. It shows why resistant mechanisms to treatment need to be elucidated. MicroRNA (miR) are short RNA, implicated in messenger ribonucleic acid (mRNA) regulation. Evidence is emerging that miR is implicated in prostate cancer response to treatment. It would be interesting to determine if a miR profile can predict treatment response to chemotherapy and/or to novel hormonal agents.

DETAILED DESCRIPTION:
Several drugs are available for metastatic castration resistant prostate cancer such as chemotherapy (docetaxel, cabazitaxel) and novel hormonal agents (abiraterone, enzalutamide), in France. The oncologist has to choose between those two type of treatment, without any biological predictor of efficacy for his patient. It is always difficult to choose knowing that 30 to 50% of patients won't benefit from the treatment chosen. It shows why resistant mechanisms to treatment need to be elucidated. MicroRNA (miR) are short RNA, implicated in messenger ribonucleic acid (mRNA) regulation. Evidence is emerging that miR is implicated in prostate cancer response to treatment. It would be interesting to determine if a miR profile can predict treatment response to chemotherapy and/or to novel hormonal agents.

ELIGIBILITY:
Inclusion Criteria:

* prostate adenocarcinoma
* metastatic disease, proven (CT or bone scintigraphy or MRI or positron emission tomography(PET)-CT or X ray)
* castration resistance, proven with biology or radiologic progression
* affiliated to a french social security regimen

Exclusion Criteria:

* other cancer within five years
* any judiciary protection measure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate cancer only concerns male people
Enrollment: 33 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
miRNA and chemotherapy | 30 months
  miRNA expression profile predicting resistance to chemotherapy
miRNA and novel hormonal agent (NHA) | 30 months
  miRNA expression profile predicting resistance to novel hormonal agents

SECONDARY OUTCOMES:
miRNA and progression free survival (PFS) | 30 months
  correlation between miRNA profile and progression free survival
miRNA and overall survival (OS) | 30 months
  correlation between miRNA profile and overall survival
miRNA in tissue sample | 30 months
  comparison between miRNA expression in serum and in tumoral tissue

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde CANCEL, MD, Study Director — University Hospital, Tours
Locations (1):
- University Hospital of Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang X, Yuan T, Liang M, Du M, Xia S, Dittmar R, Wang D, See W, Costello BA, Quevedo F, Tan W, Nandy D, Bevan GH, Longenbach S, Sun Z, Lu Y, Wang T, Thibodeau SN, Boardman L, Kohli M, Wang L. Exosomal miR-1290 and miR-375 as prognostic markers in castration-resistant prostate cancer. Eur Urol. 2015 Jan;67(1):33-41. doi: 10.1016/j.eururo.2014.07.035. Epub 2014 Aug 14. PMID 25129854
- [Background] Razdan A, de Souza P, Roberts TL. Role of MicroRNAs in Treatment Response in Prostate Cancer. Curr Cancer Drug Targets. 2018;18(10):929-944. doi: 10.2174/1568009618666180315160125. PMID 29644941
- [Background] Lin HM, Castillo L, Mahon KL, Chiam K, Lee BY, Nguyen Q, Boyer MJ, Stockler MR, Pavlakis N, Marx G, Mallesara G, Gurney H, Clark SJ, Swarbrick A, Daly RJ, Horvath LG. Circulating microRNAs are associated with docetaxel chemotherapy outcome in castration-resistant prostate cancer. Br J Cancer. 2014 May 13;110(10):2462-71. doi: 10.1038/bjc.2014.181. Epub 2014 Apr 8. PMID 24714754
- [Background] Zhang G, Tian X, Li Y, Wang Z, Li X, Zhu C. miR-27b and miR-34a enhance docetaxel sensitivity of prostate cancer cells through inhibiting epithelial-to-mesenchymal transition by targeting ZEB1. Biomed Pharmacother. 2018 Jan;97:736-744. doi: 10.1016/j.biopha.2017.10.163. Epub 2017 Nov 6. PMID 29102917
- [Background] Fletcher CE, Sulpice E, Combe S, Shibakawa A, Leach DA, Hamilton MP, Chrysostomou SL, Sharp A, Welti J, Yuan W, Dart DA, Knight E, Ning J, Francis JC, Kounatidou EE, Gaughan L, Swain A, Lupold SE, de Bono JS, McGuire SE, Gidrol X, Bevan CL. Androgen receptor-modulatory microRNAs provide insight into therapy resistance and therapeutic targets in advanced prostate cancer. Oncogene. 2019 Jul;38(28):5700-5724. doi: 10.1038/s41388-019-0823-5. Epub 2019 May 1. PMID 31043708